CLINICAL TRIAL: NCT04784637
Title: Adaptive Biobehavioral Control (ABC) of Automated Insulin Delivery: A Randomized, Controlled Pilot Study
Brief Title: Adaptive Biobehavioral Control (ABC) of Automated Insulin Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sue Brown, Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200336; 2R01DK085623-10 (NIH)
Record Dates: First submitted 2020-12-16; First posted 2021-03-05 (Actual); Results first posted 2022-12-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas (AP); Continuous Glucose Monitor (CGM); Closed Loop Control (CLC); Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insemination, Artificial, Heterologous; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Group 1 (Experimental): AID + Auto Titration Module (ATM) and Web Simulation Tool (WST) for 6 weeks
  Interventions: Device: Web Simulation Tool (WST); Device: Auto Titration Module (ATM); Device: Automated Insulin Delivery (AID) System
- Group 2 (Experimental): AID + Auto Titration Module (ATM) and Web Simulation Tool (WST) +Behavioral Adaptation Module (BAM) for 6 weeks
  Interventions: Device: Web Simulation Tool (WST); Device: Behavioral Adaptation Module (BAM); Device: Auto Titration Module (ATM); Device: Automated Insulin Delivery (AID) System

INTERVENTIONS:
Device: Web Simulation Tool (WST) — WST will allow users of the Control-IQ system replay treatment scenarios in computer simulation, thereby allowing user training with carbohydrate and insulin action.
Device: Behavioral Adaptation Module (BAM) — BAM provides on-demand information to the participant primarily on glycemic risks.
  Arms: Group 2
Device: Auto Titration Module (ATM) — ATM provides recommendations to the participant to periodically update insulin parameters.
Device: Automated Insulin Delivery (AID) System — The t:slim X2 insulin pump with Control-IQ technology, Tandem Diabetes Care will be the AID in this study.

SUMMARY:
The purpose of this pilot study is to test the safety and feasibility of using two or three research modules in conjunction with an automated insulin delivery device (AID).

DETAILED DESCRIPTION:
This concept is implemented in the Adaptive Biobehavioral Control (ABC) system - ABC will use human-machine co-adaptation of AID, recognizing both the necessity for the control algorithm to adapt to changes in human physiology, and the necessity for the person to adapt to AID action. ABC will be implemented on the Web Information Tool (WIT) platform/system and includes the following modules to be used alongside the automated insulin delivery device facilitating behavioral adaptation:

* Behavioral Adaptation Module (BAM) - a behavioral intervention deployed in a mobile app to assist a person's adaptation to automated insulin delivery by information and risk assessment primarily regarding glycemic risks, and
* Auto Titration Module (ATM) - a web-based tool with an automated procedure to track risk status and changes in the participant's metabolic profile. This module will present updated insulin control parameters to the user once a week using a web-based format accessible to the participant.
* Web-based Simulation Tool (WST) --a web-based education tool for participants to interact with their data to visualize and replay various scenarios to understand the impact of insulin parameter changes.

Design: Two-week baseline use of personal AID system followed by randomization 1:1 into two groups.

* Group 1 will use their personal AID system and add an auto titration module (ATM) and web simulation tool (WST) in which insulin parameters may be adjusted on a weekly basis.
* Group 2 will use their personal AID system and add the ATM / WST on a weekly basis as well as a behavioral adaptation module (BAM). The BAM will consist of information modules in which information only is given to participants (e.g. hypoglycemic risks).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 and ≤70 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using insulin pump for at least six months
4. Currently using insulin for at least six months
5. Currently using or anticipated to be using the t:slim X2 insulin pump with Control-IQ technology at the start of the run-in phase (Visit 1).
6. Using or willing to use insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
7. Access to internet and willingness to upload data during the study as needed
8. Willing to use an app on a smart phone during the study.
9. For females, not currently known to be pregnant or breastfeeding
10. If female, sexually active, and of childbearing potential, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
11. Willingness to use only insulin analogs approved for use in the t:slim X2 pump such as lispro (Humalog) or aspart (Novolog) and not use ultra-rapid acting insulin analogs (e.g. FiAsp) during the study
12. Total daily insulin dose (TDD) at least 10 units per day
13. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, biguanides, and sulfonylureas)
14. An understanding and willingness to follow the protocol and signed informed consent

Exclusion Criteria:

1. Concurrent use of any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas)
2. A condition, which in the opinion of the investigator or designee, would put the participant at risk or interfere with the completion of the protocol.
3. History of diabetic ketoacidosis (DKA) in the 12 months prior to enrollment
4. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
5. Currently being treated for a seizure disorder
6. Hemophilia or any other bleeding disorder
7. Planned surgery during study duration
8. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
9. Having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (e.g. study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally, data will be made available after the primary publications of each study.
Access Criteria: The Data Sharing Agreements will be formulated by the study team.

REFERENCES:
- [Background] Colmegna P, McFadden R, Fabris C, Lobo B, Nass R, Oliveri MC, Brown SA, Kovatchev B. Adaptive Biobehavioral Control: A Pilot Analysis of Human-Machine Coadaptation in Type 1 Diabetes. Diabetes Technol Ther. 2024 Sep;26(9):644-651. doi: 10.1089/dia.2023.0399. Epub 2024 Apr 30. PMID 38662425

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants signed a consent which was defined as enrollment in the protocol. 1 participant withdrew after signing the consent due to personal scheduling issues and 30 participants were randomized and reported in study results.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 38 (16) | 40 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 14 | 26
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Total Daily Insulin [Mean (Standard Deviation); unit: units per day] | 47.6 (29.9) | 45.6 (19.8) | 46.6 (24.9)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 23 (13) | 23 (15) | 23 (14)

OUTCOME MEASURES:

1. Primary Outcome: Number of SAE or ADE Related to the Use of ATM / WST and BAM Modules.
Description: Safety assessment of ATM / WST and BAM modules by assessing serious adverse events or adverse device effects deemed related to the use of ATM/WST and BAM modules specifically.
Time Frame: 6 weeks
Measure: Number; unit: events
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 15 | 15
events | 0 | 0

2. Secondary Outcome: Time in Range
Description: Percent of CGM readings in the target ranges of 70-180mg/dL from 2 weeks of baseline compared to last 2 weeks of treatment period.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Group 1 Baseline Measure: Two-week of baseline measures.
- Group 1 Post Randomization: AID + Auto Titration Module (ATM) and Web Simulation Tool (WST) for 6 weeks
  Web Simulation Tool (WST): WST will allow users of the Control-IQ system replay treatment scenarios in computer simulation, thereby allowing user training with carbohydrate and insulin action.
  Auto Titration Module (ATM): ATM provides recommendations to the participant to periodically update insulin parameters.
  Automated Insulin Delivery (AID) System: The t:slim X2 insulin pump with Control-IQ technology, Tandem Diabetes Care will be the AID in this study.
- Group 2 Baseline: Two weeks of baseline measures
- Group 2 Post Randomization: AID + Auto Titration Module (ATM) and Web Simulation Tool (WST) +Behavioral Adaptation Module (BAM) for 6 weeks
  Web Simulation Tool (WST): WST will allow users of the Control-IQ system replay treatment scenarios in computer simulation, thereby allowing user training with carbohydrate and insulin action.
  Behavioral Adaptation Module (BAM): BAM provides on-demand information to the participant primarily on glycemic risks.
  Auto Titration Module (ATM): ATM provides recommendations to the participant to periodically update insulin parameters.
  Automated Insulin Delivery (AID) System: The t:slim X2 insulin pump with Control-IQ technology, Tandem Diabetes Care will be the AID in this study.
Arm/Group | Group 1 Baseline Measure | Group 1 Post Randomization | Group 2 Baseline | Group 2 Post Randomization
Number analyzed (Participants) | 15 | 15 | 15 | 15
percentage of time | 77.0 (11.6) | 73.8 (8.1) | 74.6 (9.4) | 74.6 (8.9)
Statistical Analysis 1: Comparison: Group 1 Baseline Measure vs Group 1 Post Randomization; Test type: Superiority; p = 0.064, t-test, 2 sided
Statistical Analysis 2: Comparison: Group 2 Baseline vs Group 2 Post Randomization; Test type: Superiority; p = 0.97, t-test, 2 sided

3. Secondary Outcome: Time in Hypoglycemia
Description: Percent of CGM readings <70 mg/dL
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Group 1 Baseline Measure | Group 1 Post Randomization | Group 2 Baseline | Group 2 Post Randomization
Number analyzed (Participants) | 15 | 15 | 15 | 15
percentage of time | 2.35 (1.98) | 1.41 (1.33) | 1.58 (1.71) | 1.48 (1.30)
Statistical Analysis 1: Comparison: Group 1 Baseline Measure vs Group 1 Post Randomization; Test type: Superiority; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Group 2 Baseline vs Group 2 Post Randomization; Test type: Superiority; p = 0.93, t-test, 2 sided

4. Secondary Outcome: INSPIRE Questionnaire
Description: Questionnaire addressing system/technology use. The INSPIRE questionnaire assesses user expectations and experiences with Insulin Delivery Systems: Perceptions, Ideas, Reflections, Expectations (INSPIRE). Survey total scores are computed by calculating the mean of the sum of all item ratings then multiplying the mean by 25 to scale the score to a range from 0 to 100. Higher scores indicate a more positive perception of insulin delivery systems. Items are rated on a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The Adult survey has 22 items.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 Baseline Measure | Group 1 Post Randomization | Group 2 Baseline | Group 2 Post Randomization
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale | 77 (12) | 74 (8) | 75 (9) | 75 (9)

ADVERSE EVENTS:
Time Frame: Duration of study which was approximately 8 weeks.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT04784637/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT04784637/ICF_001.pdf